CLINICAL TRIAL: NCT02846493
Title: Efficacy and Safety of Dexamethasone Prevention for Patients of Ovarian Hyperstimulation Syndrome -- A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Efficacy and Safety of Dexamethasone Prevention for Patients of Ovarian Hyperstimulation Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-ohss-001
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Ovarian hyperstimulation syndrome; Dexamethasone
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Bromocriptine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bromocriptine group (Active Comparator): Rectal bromocriptine (2.5 mg, qd) for 7 days
  Interventions: Drug: bromocriptine
- dexamethasone group (Experimental): Oral take dexamethasone(3mg,qd)for 7 days
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: bromocriptine — Patients in this group will receive rectal bromocriptine at a daily dose of 2.5 mg for 7 days,from the day of oocyte pickup.At oocyte retrieval and at the 3rd d and 5th d of treatment, all the patients received the measurements of body mass index (BMI), abdominal circumference (AC), maximum depth of ascites in ultrasonic (D),hepatorenal function, coagulation function ,white blood cell count (WBC), hematocrit (HCT), Vascular Endothelial Growth Factor(VEGF),drink intake (Intake) and urine volume.
  Arms: bromocriptine group
Drug: dexamethasone — Patients in this group will take oral dexamethasone at a daily dose of 3mg for 7 days,from the day of oocyte pickup.At oocyte retrieval and at the 3rd d and 5th d of treatment, all the patients received the measurements of body mass index (BMI), abdominal circumference (AC), maximum depth of ascites in ultrasonic (D),hepatorenal function, coagulation function ,white blood cell count (WBC), hematocrit (HCT),Vascular Endothelial Growth Factor(VEGF), drink intake (Intake) and urine volume.
  Arms: dexamethasone group

SUMMARY:
This prospective, randomized, controlled clinical trial will evaluate the effect and security of dexamethasone prevention for Patients of Ovarian Hyperstimulation Syndrome.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is a iatrogenic complication of ovarian stimulation,which in its severe form is associated with significant morbidity and can be life threatening. It is characterized by cystic enlargement of the ovaries and rapid fluid shifts from the intravascular compartment to the third space. It is thought that increased vascular permeability is the pivotal mechanism of OHSS pathophysiology. The administration of human chorionic gonadotrophin results in the release of vasoactive substance such as vascular endothelial growth factor that causes vasodilation and leakage of fluids. Glucocorticoids and their synthetic derivatives have an inhibitory effect on the VEGF gene expression in vascular smooth muscle cells. By reducing leukocytic infiltration and the release of inflammatory mediator, inhibiting vasodilation and preventing increases in vascular permeability, these agents can dampen the inflammatory response and prevent edema formation ,thus offering a potential therapeutic intervention for OHSS. Investigators have observed more than a hundred patients in clinical practice that low-dose dexamethasone has prevention action for patients in IVF cycles at high risk of OHSS. This clinical trial is designed to evaluate the effect and security of dexamethasone prevention for patients of Ovarian Hyperstimulation Syndrome. There are two groups: bromocriptine group, dexamethasone group .After followed-up for 7 days , Clinical OHSS parameters will be collected at oocyte retrieval and at the 4rd d and 6th d of treatment .

ELIGIBILITY:
* Inclusion Criteria:

  * Women of reproductive age
  * Women having controlled ovarian hyperstimulation as part of any assisted reproductive technique
  * Women at risk of severe OHSS(serum estradiol levels were>3000pg/ml on the day of HCG trigger ; there was retrieval of 20 or more oocytes)
* Exclusion Criteria:

  * Unwillingness to comply with the study protocol.
  * Attending other clinical trials in the same period.
  * Chronic glucocorticoid their synthetic derivatives intake.
  * History of allergic to study medications.
  * The patients who cannot take dexamethasone.： hypertension, diabetes,gastric ulcer; abnormal renal or hepatic function and so on.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate and severe OHSS | 7 days
  Moderate OHSS is characterized by the presence of ascites on ultrasound examination ,moderate hemoconcentration and elevated leukocytes.Symptoms include abdominal distension , nausea and vomiting . And diagnosis of severe OHSS required clinical evidence of ascites or hydrothorax or breathing difficulties or one of the following criteria: 1) increased blood viscosity i.e. hemoglobin at least 15 gm%, hematocrit at least 45%, or leucocyte count at least 20,000 per cubic millimeter. 2) coagulation abnormality.3) liver dysfunction, defined when transaminases (AST or ALT) are more than 40 u/ml.

SECONDARY OUTCOMES:
Adverse side effects of treatment | 7 days
  Number of participants with treatment-related adverse events as assessed by CTCAE V4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zeng, Principal Investigator — Reproductive medicine center , 6th Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Sixth Affiliated Hospital,Sun Yat-Sen University, Guangzhou, Guangdong, China